CLINICAL TRIAL: NCT02928705
Title: Comparison of Analgesic Treatment Quality Between Prehospital Emergency Care of Telemedically Guided Paramedics and On-scene Physicians - a Retrospective Longitudinal Study
Brief Title: Quality of Telemedically Guided Prehospital Analgesia
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: Quality of Tele-Analgesia
Record Dates: First submitted 2016-07-28; First posted 2016-10-10 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Analgesia; Prehospital; Telemedicine; Ambulance; Opioids; Teleconsultation; Tele-emergency Medical Services; Adverse Events; City of Aachen; Prehospital Emergency Medical Service Physician
Keywords: analgesia; prehospital; telemedicine; ambulance; opioids; teleconsultation; tele-emergency medical services; adverse events; prehospital emergency medical service physician
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- telemedicine group: physician operated telemedical prehospital analgesia
  Interventions: Procedure: physician operated telemedical prehospital analgesia
- historical control group: prehospital analgesia by on-scene EMS physicians
  Interventions: Procedure: prehospital analgesia by on-scene EMS physicians

INTERVENTIONS:
Procedure: physician operated telemedical prehospital analgesia — Ambulances in the EMS of the city of Aachen are equipped with a portable telemedicine system. In emergencies requiring intravenous analgesia paramedics can use this system to contact the tele-EMS physician with an audio-connection. Vital parameters (e.g., ECG, pulse oximetry, non-invasive blood pressure) can be transferred in real-time. The transmission of still pictures - taken with an official smartphone - and video streaming from the inside of the ambulance are also possible. The tele-EMS physician supports the paramedics and can delegate the application of morphine and other analgesics based on two predefined algorithms for trauma and non-trauma cases that are displayed on a context-sensitive telemedical documentation system in the teleconsultation center.
  Groups: telemedicine group
Procedure: prehospital analgesia by on-scene EMS physicians — This (control) group represents the conventional treatment in German emergency medical service (EMS). In addition to an ambulance manned with paramedics, a prehospital EMS physician is deployed to conduct analgesic treatment on-scene. Treatment data for this group are selected from the time period before implementing teleconsultation in routine and therefore represent a historical control group.
  Groups: historical control group

SUMMARY:
The purpose of this retrospective study is to analyze quality and adverse events of analgesia by telemedically supported paramedics in comparison to conventional treatment by on-scene emergency medical service (EMS) physicians in the EMS of the city of Aachen, Germany.

DETAILED DESCRIPTION:
The standard emergency medical service (EMS) in Germany consists of a two-tiered system with ambulances (paramedics) and prehospital EMS physician units. For example, legal conditions restrict opioid-based analgesia to physicians. Based on pre-defined standards regional emergency dispatch centers deploy both kinds of emergency units.

In recent years telemedicine emerged as a complementary system in EMS that may provide remote medical expertise and sustain or even improve quality of medical treatment on-scene. Particularly, based on the results of the projects Med-on-@ix and TemRas (telemedical rescue assistance system), emergency telemedical services were gradually implemented in daily routine of the EMS of the city of Aachen, Germany.

In this retrospective study the quality and adverse events of analgesia by telemedically supported paramedics shall be compared to conventional treatment by on-scene EMS physicians in the EMS of the city of Aachen, Germany.

ELIGIBILITY:
Inclusion Criteria:

* Initial Numerical Rating Scale ≥ 5 and
* Documented administration of analgesics

Exclusion Criteria:

* Missing consent for telemedical consultation (in teleconsultation group)
* Initial NRS < 5
* Analgesia in non-ST-segment elevation acute coronary syndrome (Non-STEMI-ACS) and ST-elevating myocardial infarction (STEMI)
* Initially unconscious patient
* Inter-hospital transfer missions
* Cases involving both on-scene and telemedical-EMS physicians

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients requiring prehospital pain treatment in the EMS of the city of Aachen
Sampling Method: Probability Sample
Enrollment: 381 (Actual)
Dates: Start 2014-01; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Quality of analgesia | Time span of the respective prehospital emergency case treatment; on average a time interval of 30 - 120 minutes for each case.
  Decrease of value on the Numerical Rating Scale (NRS; 0-10). The NRS is applied at initial contact with the patient and at the end of the mission.

SECONDARY OUTCOMES:
Rate of adverse events | Time span of the respective prehospital emergency case treatment; on average a time interval of 30 - 120 minutes for each case.
  Respiratory and/or circulatory insufficiency and/or severe allergic reactions
Administered analgesics and their dosages | Time span of the respective prehospital emergency case treatment; on average a time interval of 30 - 120 minutes for each case.
Number of patients with documented analgesia related (safety-) parameters (evaluated for each safety parameter separately) | Time span of the respective prehospital emergency case treatment; on average a time interval of 30 - 120 minutes for each case.
  Documentation of analgesia related parameters:
  heart rate (beats per minute), blood pressure (mmHg), oxygen saturation (0-100%), respiratory rate (respirations per minute), Glasgow coma scale (Numerical values 3 to 15), The above named parameters should be documented by EMS teams at first medical contact and at patient handover in the emergency room.
Occurrence of nausea and vomiting | Time span of the respective prehospital emergency case treatment; on average a time interval of 30 - 120 minutes for each case.

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Rossaint, Professor, MD, Study Chair — University Hospital, Aachen; Sebastian Bergrath, MD, Principal Investigator — University Hospital, Aachen
Locations (1):
- University Hospital Aachen, Aachen, Germany

IPD SHARING:
Plan to Share IPD: No
No additional research benefits.